CLINICAL TRIAL: NCT02845388
Title: Sildenafil Citrate for Endometrial Preparation in Frozen-thawed Embryo Transfer Cycles
Brief Title: Sildenafil Citrate in Frozen Embryo Transfer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omar Ahmed El Sayed Saad (Other)
Responsible Party: Sponsor-Investigator, Omar Ahmed El Sayed Saad, Resident of obstetric and gynecology in Shebin Elkom teaching hospital, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ainshams2015Omar
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
Keywords: IVF
MeSH Terms: conditions — Infertility | interventions — Sildenafil Citrate; Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- estradiol valerate (Active Comparator): estradiol valerate 2mg every 12 hours orally starting from the second day of the menstrual cycle till reaching trilaminar endometrial pattern and endometrial thickness 8 mm or more
  Interventions: Drug: estradiol valerate
- Sildenafil citrate and estradiol valerate (Active Comparator): Sildenafil citrate 25 mg every 6 hours orally in combination with estradiol valerate 2mg every 12 hours orally starting from the second day of the menstrual cycle till reaching trilaminar endometrial pattern and endometrial thickness 8 mm or more
  Interventions: Drug: Sildenafil citrate; Drug: estradiol valerate

INTERVENTIONS:
Drug: Sildenafil citrate
  Other Names: Viagra
  Arms: Sildenafil citrate and estradiol valerate
Drug: estradiol valerate

SUMMARY:
Comparison between usage of Sildenafil citrate with estradiol valerate or estradiol valerate alone in endometrial preparation and outcome of frozen-thawed embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

* all cases have at least 2 good quality blastocysts available for transfer

Exclusion Criteria:

* uterine structural abnormalities
* advanced uterine disease
* hydrosalpinx and pyosalpinx

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
endometrial pattern | starting from 8th day till 12th day of the menstrual cycle
  Endometrial pattern will be trilaminar or bilaminar after it's preparation with estradiol valerate alone or estradiol valerate and sildenafil citrate. Endometrial pattern will be estimated by transvaginal ultrasonography for trilaminar pattern every other day from 8th day till 12th day of the menstrual cycle.

SECONDARY OUTCOMES:
endometrial thickness | starting from 8th day till 12th day of menstrual cycle
  Endometrial thickness will be estimated by transvaginal ultrasonography after it's preparation with estradiol valerate alone or estradiol valerate and sildenafil citrate for thickness 8 mm or more every other day from 8th day till 12th day of the menstrual cycle.
biochemical pregnancy test | 2 weeks after embryo transfer
  Serum B,human chorionic gonadotropin subunit will be measured 2 weeks after embryo transfer which will be positive when it's level exceeds 5 milli international unit /milli litre in patient's serum.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa mohamed elghannam, professor, Study Chair — department of obstetric and gynacology Ain shams university

IPD SHARING:
Plan to Share IPD: Yes